CLINICAL TRIAL: NCT05117346
Title: An Exploratory Safety and Efficacy Clinical Study of CARDIX-101 for the Treatment of Chronic Bradycardia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardix Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CARDIX Therapeutics LLC
Record Dates: First submitted 2021-10-24; First posted 2021-11-11 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Intervention Model Description: The study investigates three dosage levels of CARDIX-101 (CARDIX-101A, CARDIX-101B, and CARDIX-101C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- To Establish the Safety and Efficacy of CARDIX-101 in Chronic Bradycardia Patients (Experimental): Treatment Regimen: A total of 20±4 chronic bradycardia subjects with a heart rate (H.R.) average of less than 60 bpm will be enrolled in the study (6±3/cohort). A clinical study period of 14±2-days is planned for each enrollment of patients.
  Route of Administration: Each subject will receive, via oral administration, one capsule of study medicine per dose and three doses per day for 14±2-days treatment.
  Interventions: Drug: CARDIX-101A, CARDIX-101B, CARDIX-101C

INTERVENTIONS:
Drug: CARDIX-101A, CARDIX-101B, CARDIX-101C — Each subject will receive, via oral administration, one capsule of study medicine per dose and three doses per day for 14±2-days treatment.
  Other Names: CARDIX-101

SUMMARY:
The treatment of chronic bradycardia, one of the cardiovascular diseases, remains an essential unsolved issue. The objective of this project is to speed up a new drug CARDIX-101 clinical Phase 1IA trial for the treatment of chronic bradycardia and to solve an unmet medical need.

To date, there is no regulatory approved drug of this type available in the U.S or the world. If the new drug CARDIX-101 demonstrated a significant positive effect on chronic bradycardia, it should have a sizeable demand and solve an unmet medical need.

DETAILED DESCRIPTION:
Following FDA and ICH Good Clinical Practice (GCP) guidance, a clinical Phase I study titled "A Single Ascending Dose Clinical Study to Establish Safety and Tolerability of CARDIX-101 in Bradycardia Patients" was conducted at the University of California San Diego (UCSD) School of Medicine, Cardiac Electrophysiology Center, and Altman Clinical and Translational Research Institute and was completed in August 2020 under IND# 131775.

The clinical Phase 1 study of CARDIX-101 was completed using eighteen patients with six ascending single-dose levels. There were no adverse effects observed or reported for all participating subjects related to the investigational medicine.

A current clinical Phase IIA study, "An Exploratory Safety and Efficacy Study of CARDIX-101 for the treatment of Chronic Bradycardia," is a multi-center clinical study. The current clinical study is designed to utilize appropriate wearable monitoring devices for today's Decentralized Clinical Trial.

This study will consist of a multi-site clinical exploratory study in chronic bradycardia patients. The study is open-label, and enrollment of a cohort occurs without randomization.

The study investigates three dosage levels of CARDIX-101 (CARDIX-101A, CARDIX-101B, and CARDIX-101C). The initial cohort will be enrolled in a staggered manner. In this way, it will make the clinical study more accessible for the patient to participate.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has bradycardia (H.R. <60 BPM). The subject's symptoms, if any, such as dizziness, confusion, fatigue, shortness of breath, chest pain, and syncope, are required to be documented in the case report form (CRF) in the screening, treatment, and follow-up periods.
2. The subject has been informed of the investigational nature of this study and has completed a written informed consent form (ICF) in accordance with institutional, local, and national guidelines.
3. The subject is able to return for the safety and efficacy follow up period and provides at least two modes of contact information (e.g., home and mobile phone numbers, address) and contact information for at least one close contact (e.g., family member or friend) to facilitate follow up.
4. The subject is a male or female 18-80 years of age.

Exclusion Criteria:

1. Patients with peptic ulcer disease, seizure disorder, or cardiac arrhythmia with tachycardia are excluded
2. Patients with asthma who are already taking a beta-agonist and/or Theophylline are excluded
3. Pregnancy (all women of childbearing potential, unless surgically sterilized or post-menopausal defined as the cessation of menses for over one year, receive a pregnancy test).
4. Systolic blood pressure is <100 mmHg.
5. Heart rate >60 bpm.
6. Severe bradycardia or sinus pauses, which in the opinion of the P.I. requires urgent pacemaker implantation or A.V. block > 2nd degree, or existing implanted pacemaker.
7. Serum potassium <4.0 mEq/L or mmol/L by the local laboratory at the screening.
8. History of receiving another Class I or Class III antiarrhythmic drug within three days prior to enrollment. Excluded Class I antiarrhythmic drugs include quinidine, procainamide, disopyramide, lignocaine, mexiletine, flecainide, and propafenone. Excluded Class III drugs include dofetilide, sotalol, dronedarone, and ranolazine.
9. There is a history of amiodarone (oral or IV) within 90 days prior to the study.
10. There is native or prosthetic aortic or mitral stenosis with aortic valve area ≤1.0 cm2, or mitral valve area of <1.5 cm2 or any other valvular diseases requiring surgery.
11. There is an ejection fraction of <35% within one year prior to enrollment (most recent measure if more than one).
12. Atrial fibrillation (A.F.) or atrial flutter (AFL) as a result of surgery (postoperative AF/AFL) within 30 days prior to the study.
13. There is a history of electrical cardioversion within seven calendar days prior to the study.
14. There is a history of any polymorphic ventricular tachycardia, including torsade de points.
15. History or family history of long Q.T. syndrome or other inherited arrhythmia syndrome.
16. There is a history of ventricular tachycardia requiring drug or device therapy.
17. Participation in another investigational drug or device trial within 30 days prior to the study. (subjects in registries may participate with the approval of the registry sponsor.)
18. Acute cardiovascular events (myocardial infarction, pulmonary embolism, cerebrovascular accident, unstable angina, or transient ischemic attack) within 90 days prior to enrollment.
19. Psychiatric disorder, active alcohol/drug abuse, or other circumstance or condition that, in the Investigator's opinion, may interfere with any aspect of protocol adherence or a subject's ability to give informed consent.
20. Untreated hyperthyroidism or hypothyroidism.
21. Acute pericarditis.
22. Unrelated illness such as substantial infection, fever, or prescribed antibiotics in the last seven days, acute rheumatic fever, metastatic cancer, severe hepatic disease, or other extreme medical conditions
23. Exclusion of a woman who is breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint | The time frame is during medication 14±2 days
  The primary endpoint measures the mean Heart Rate.
  During the treatment period of 14±2-day, each patient is required to use near-real-time HR/ECG monitoring for a total of 14±2-day with no less than 16±6-hours of monitoring per day.
  The increase in the clinical study period (14±2 days) for a patient compared to patient heart rate before dosing of CARDIX-101 (either by baseline record for 2-hours or historical patient records for mean Heart Rate of 5-days).
  The measure results are as follows:
  Effectiveness/Significance Level 1: H.R. increase 5-10% Effectiveness/Significance Level 2: H.R. increase 10-15% Effectiveness/Significance Level 3: H.R. increase 15-20% Effectiveness/Significance Level 4: H.R. increase ≥20%

CONTACTS AND LOCATIONS:
Locations (1):
- SpaceMed-X, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to make individual participant data available to other research.